CLINICAL TRIAL: NCT03693482
Title: The Validity and Reliability of the Four Square Step Test in Typically Developed Children
Brief Title: The Validity and Reliability of the Four Square Step Test
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Emine Handan Tüzün, Professor, Eastern Mediterranean University
Other Study IDs: ETK00-2018-0202
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Only Child; Balance, Postural

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: the Four Square Step test — A square will be formed by using four 90 cm long canes placed on the ground. The sequence will be explained and demonstrated to the participants. They will be allowed one practice trial and subsequently two trials. Instructions will be given and encouraged to complete the sequence as fast as possible without touching the canes. The sequence of trial was 1,2,3,4,1,4,3,2,1. If a participant touch the canes, or perform the test sequence inaccurately, or both feet of the participant do not make contact with the floor in each square, the trial will be considered as unsuccessful and the test will be repeated. One unsuccessful trial will be allowed. The best time will be taken as the score of FSST which are completed successfully.

SUMMARY:
This study will evaluate concurrent and discriminative validity, reliability and level of agreement between the Timed Up & Go test and the four square step test in typically developed children.

DETAILED DESCRIPTION:
Participants will be assessed by two physiotherapists on two separate days. Prior to the trial, testing instructions to be delivered to participants will be translated and adapted into Turkish. In order to maximize potential agreement and to improve rating accuracy, reliability, and validity, assessment skills of the raters will be refreshed through training.

Administration of the tests will be performed in a corridor of the school. Assessments will be performed in a quiet and adequately lighted environment to minimize the distraction. Participants will be tested with their regular footwear. The demographic information of participants will be recorded. The dynamic balance performances on the four square step test (FSST) and the Timed up & Go test (TUG) will be assessed by Rater A and B independently and these assessments repeated 24-h later. The participants will be allowed to rest up to five minutes between sessions. A stopwatch will be used to measure time to complete the FSST and TUG test.

Evaluations of concurrent and discriminative validity will be based on mean scores from the first measurement of rater A. Pearson's correlation coefficient (r) will be used to assess the concurrent validity of the FSST and TUG tests. Between-groups discriminative validity of the FSST will be evaluated by the one-way analysis of variance (ANOVA) with Bonferroni post-hoc test. Both intra- and inter-rater reliability will be assessed using intraclass correlation coefficients (ICC). ICC2,1 and ICC2,2 estimates and their 95% confidence intervals will be calculated based on absolute-agreement. Bland & Altman plots will be constructed to demonstrate agreement between TUG and FSST, and between assessments of rater A and B.

ELIGIBILITY:
Inclusion Criteria:

* aged 5 to 10 years,

Exclusion Criteria:

* have musculoskeletal or neurological disorders,
* have history of surgeries of the spine or orthopedic,
* have uncorrected visual acuity.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Typically developed children between the ages of 5-10 in Cihangir-Düzova Elementary School in Famagusta, North Cyprus.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
The Four Square Step test | At baseline
  Assessing of the dynamic balance in typically developed children. A square will be formed by using four 90 cm long canes placed on the ground. Instructions will be given and encouraged to complete the sequence as fast as possible without touching the canes. The sequence of trial was 1,2,3,4,1,4,3,2,1. The best time will be taken as the score of FSST which are completed successfully.

SECONDARY OUTCOMES:
The Time Up and Go test | At baseline
  Assessing of the dynamic balance in typically developed children. A three meter pathway on the testing floor will be marked with red colored masking tape. The TUG will be administered using 2 standard chairs. The best time will be taken as the score of TUG which are completed successfully.

CONTACTS AND LOCATIONS:
Overall Officials: Emine H Tüzün, Prof. PhD., Study Chair — Eastern Mediterranean University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation,; Levent Eker, Assist.Prof., Principal Investigator — Eastern Mediterranean University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation,; Selma Uzuner, MSc.,PT., Principal Investigator — Eastern Mediterranean University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation,; Buse Sezerel, MSc.,PT., Principal Investigator — Girne Akçiçek Hospital; Hayriye Tomaç, MSc.,PT., Principal Investigator — Eastern Mediterranean University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation,; Serpil Mıhçıoğlu, MSc.,PT., Principal Investigator — Eastern Mediterranean University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation,; Wayne Dite, BAppSci (PE), Principal Investigator — Austin Hospital Royal Talbot Rehabilitation Center, Kew, Vic, Australia
Locations (1):
- 1. Eastern Mediterranean University Health Sciences Faculty, Department of Physiotherapy and Rehabilitation,, Ankara, Turkey (Türkiye)